CLINICAL TRIAL: NCT05121051
Title: Phase II Randomized, Double Blind, Placebo-Controlled Trial of Broccoli Seed and Sprout Extract (BSSE), Avmacol ES, to Evaluate Sustained Detoxification of Tobacco Carcinogens in Heavy Smokers
Brief Title: Testing the Effect of the Broccoli Seed and Sprout Extract, Avmacol ES, on the Cancer Causing Substances of Tobacco in Heavy Smokers
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NCI-2021-12014; NCI-2021-12014 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00000614 (Other: University of Arizona Cancer Center - Prevention Research Clinic); UAZ21-06-01 (Other: DCP); P30CA023074 (NIH); UG1CA242596 (NIH)
Record Dates: First submitted 2021-11-13; First posted 2021-11-16 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Cigarette Smoking-Related Carcinoma
MeSH Terms: interventions — Specimen Handling

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group I (broccoli seed and sprout extract) (Experimental): Patients receive broccoli seed and sprout extract PO QD for 12 weeks in the absence of unacceptable toxicity. Patients undergo the collection of blood, nasal epithelial cell, and buccal cell samples throughout the study.
  Interventions: Procedure: Biospecimen Collection; Dietary Supplement: Broccoli Sprout/Broccoli Seed Extract Supplement; Other: Questionnaire Administration
- Group II (placebo) (Active Comparator): Patients receive placebo PO QD for 12 weeks in the absence of unacceptable toxicity. Patients undergo the collection of blood, nasal epithelial cell, and buccal cell samples throughout the study.
  Interventions: Procedure: Biospecimen Collection; Drug: Placebo Administration; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood, buccal cell, and nasal epithelial cell samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Dietary Supplement: Broccoli Sprout/Broccoli Seed Extract Supplement — Given PO
  Other Names: Avmacol
  Arms: Group I (broccoli seed and sprout extract)
Drug: Placebo Administration — Given PO
  Arms: Group II (placebo)
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II trial tests whether broccoli seed and sprout extract works to break down cancer causing substances of tobacco in heavy smokers. Smokers are at increased risk for developing lung, head and neck, and other cancers. Broccoli seed and sprout extract may help break down and remove toxic substances caused by tobacco use and possibly produce substances that may protect cells from tobacco smoke-induced damage in current smokers.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine whether broccoli sprout/broccoli seed extract supplement (broccoli seed and sprout extract [BSSE]) sustainably increases the urinary excretion of the mercapturic acids of the tobacco carcinogens benzene and/or acrolein over a 12-week exposure period in otherwise healthy, current smokers.

SECONDARY OBJECTIVES:

I. To evaluate the safety and tolerability of BSSE over a 12-week exposure period.

II. To evaluate whether BSSE sustainably increases the urinary excretion of the mercapturic acid of the tobacco carcinogen crotonaldehyde.

III. To evaluate the bioavailability of BSSE measured as sulforaphane (SF) metabolites and assess for a dose-response relationship between the effective SF dose delivered by BSSE and the detoxification of benzene and acrolein.

IV. To determine whether the GSTM1 and GSTT1 genotypes are important genetic modulators of detoxification of tobacco carcinogens in the setting of prolonged exposure to BSSE.

EXPLORATORY OBJECTIVES:

I. To evaluate modulation of mucosal signatures of nuclear factor-erythroid factor 2-related factor 2 (NRF2) activation, inflammation, and innate immunity.

II. To evaluate modulation of nasal epithelial gene signatures including smoking, lung cancer, and squamous dysplasia.

OUTLINE: Patients are randomized to 1 of 2 groups.

GROUP I: Patients receive broccoli seed and sprout extract orally (PO) once daily (QD) for 12 weeks in the absence of unacceptable toxicity. Patients undergo the collection of blood, nasal epithelial cell, and buccal cell samples throughout the study.

GROUP II: Patients receive placebo PO QD for 12 weeks in the absence of unacceptable toxicity. Patients undergo the collection of blood, nasal epithelial cell, and buccal cell samples throughout the study.

After completion of study, patients are followed up at 2-4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male or female current tobacco smokers with >= 20 pack years of self-reported smoking exposure and a current average use of >= 10 cigarettes/day
* Age >= 18 years. No upper age limit
* Karnofsky performance scale >= 70%
* Absolute neutrophil count >= 1,000/microliter
* Platelets >= 100,000/microliter
* Total bilirubin =< 2 x institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3 x ULN
* Creatinine =< 1.5 x ULN
* Participants with known human immunodeficiency virus (HIV) infection are not eligible for this trial due to potential interaction between sulforaphane and anti-retroviral therapy
* Participants with a history of hepatitis C virus (HCV) infection must have been treated and cured. Participants with HCV infection who are currently on treatment are not eligible due to potential interaction between sulforaphane and anti-retroviral therapy
* The effects of BSSE on the developing human fetus at the recommended therapeutic dose are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her study physician immediately
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* History of invasive cancer within the past 2 years, except for excised and cured non-melanoma skin cancer or carcinoma in situ of the cervix. Participants who continue adjuvant treatment for an index cancer occurring > 2 years ago, such as adjuvant hormonal therapy for breast cancer, are excluded. Participants who are on anti-neoplastic treatment for a chronic malignancy, such as multiple myeloma or chronic myelogenous leukemia, are excluded
* Ongoing use of a nutraceutical or dietary supplement containing glucoraphanin or sulforaphane

  * Note, participants will be eligible if they agree to stop the glucoraphanin or sulforaphane product at least 7 days prior to the baseline visit (7-day washout)
* Participants with known chronic hepatitis B virus (HBV) infection are not eligible for this trial due to potential interaction between sulforaphane and suppressive anti-viral therapy
* Participants may not be receiving any other investigational agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to Avmacol ES® (BSSE)
* Uncontrolled intercurrent illness including, but not limited to, serious ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia
* Any other condition or lifestyle factor, that, in the opinion of the principal investigator, may adversely affect the participant's ability to complete the study or its measures or pose significant risk to the participant
* Pregnant or lactating women. Pregnant women are excluded from this study because the effects of BSSE on the developing human fetus are unknown. Because there is an unknown but potential risk for adverse events (AEs) in nursing infants secondary to treatment of the mother with BSSE, Breastfeeding should be discontinued if the mother is treated with BSSE

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 135 (Estimated)
Dates: Start 2022-09-21 (Actual); Primary Completion 2027-01-13 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Detoxification of benzene and acrolein | At baseline and 2, 4, 8, and 12 weeks
  Measured by changes in the urinary levels of their respective mercapturic acids, SPMA and 3-HPMA, from baseline.

SECONDARY OUTCOMES:
Incidence of adverse events (AE)s | Up to 12 weeks
  Measured by National Cancer Institute Common Terminology Criteria for Adverse Events version 5. The frequency and associated percentage of each specific AE will be tabulated by the treatment group and then compared via Fisher's exact test. The tolerability will be measured by the adherence rate and will be compared between the broccoli seed and sprout extract (BSSE) and placebo groups via Fisher's exact test.
Increases in detoxification of crotonaldehyde | At baseline and 2, 4, 8, and 12 weeks
  Will determine whether BSSE sustainably increases the detoxification of crotonaldehyde, as measured by changes in the creatinine-normalized urinary levels of its mercapturic acid metabolite, 3-HMPMA, over time. Similar to the carcinogens, benzene and acrolein, the detoxification of crotonaldehyde will be measured by change at 2 weeks, 4 weeks, 8 weeks and 12 weeks in the urinary excretion of 3-HMPMA from baseline, and a linear mixed effects model will be fit to changes in log-transformed urinary 3-HMPMA levels from baseline.
Bioavailability of BSSE | At baseline and 2, 4, 8, and 12 weeks
  Measured by urinary sulforaphane (SF) metabolites.
Dose-response relationship between effective SF dose and the detoxification of benzene and acrolein | Baseline up to 12 weeks
  A dose-response relationship between SF metabolites and detoxification of benzene and/or acrolein will be assessed by a linear mixed effects model with random intercepts, in which changes from baseline in each of the log-transformed urinary mercapturic acid levels as the dependent variable (response) and changes from baseline in SF metabolites as the independent variable (dose).
Genetic modulators of detoxification of tobacco carcinogens | Up to 12 weeks
  Will assess whether the GSTM1 and GSTT1 genotypes are important genetic modulators of detoxification of tobacco carcinogens in the setting of prolonged exposure to BSSE. The association of GSTM1 and GSTT1 genotypes with detoxification of benzene and/or acrolein will be assessed by a linear mixed effects model with random intercepts for changes from baseline in each of the log transformed mercapturic acid levels, in which the fixed effects include BSSE, genotype and time indicators and two-way and three-way interactions of BSSE, genotype and time indicators. This will allow us to study whether 1) the BSSE effect if significant is modulated by the genotypes, 2) the time effect if significant is modulated by the genotypes, or 3) the interaction effect between BSSE and time if significant is modulated by the genotypes.

OTHER OUTCOMES:
Change in mucosal signatures of NRF2 activation, inflammation, and innate immunity | Baseline up to 12 weeks
  Measured by the NanoString nCounter® PanCancer panel.
Modulation of nasal epithelial gene signatures | Up to 12 weeks
  Will assess modulation of nasal epithelial gene signatures including smoking, lung cancer, and squamous dysplasia.

CONTACTS AND LOCATIONS:
Overall Officials: Julie E Bauman, Principal Investigator — George Washington University Cancer Center
Locations (3):
- United States (3):
  - University of Arizona Cancer Center - Prevention Research Clinic, Tucson, Arizona
  - George Washington University Medical Center, Washington D.C., District of Columbia
  - Roswell Park Cancer Institute, Buffalo, New York

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm